CLINICAL TRIAL: NCT06294080
Title: The Effects of Eight-week Dance and Tai Chi on Balance, Well-being and Mood Among Healthy Adults
Brief Title: Effects of Dance and Tai Chi on Balance and Wellbeing on Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wolverhampton (Other)
Responsible Party: Principal Investigator, Matthew Wyon, Professor Exercise Physiology, University of Wolverhampton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DfH2023
Record Dates: First submitted 2024-01-23; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: General Population
Keywords: Balance; Well-being; Leg strength; Mood
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Random Controlled Trial: Blind
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collection carried out by RAs blinded to participants' group allocation Statistician blinded to the group and test parameters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dance (Experimental): Participants will be provided with three dance genre options to choose from, ballroom dance, street dance/Hip-pop and ballet, and the most-voted genre will be delivered. Dance sessions are instructed twice a week for eight weeks. Every session lasts 45-60 minutes, containing 5-10 minutes of warm-up and 35-55 minutes of learning or practicing. In the first four weeks, a short dance sequence will be taught and in the following four weeks, participants will mainly practicing the learnt sequence along with music.
  Interventions: Other: Dance
- Tai Chi (Experimental): The Tai Chi Group will be given the essential 18-form of Chen's style Tai Chi Chuan. Each session lasts 45-60 minutes, twice a week for 8 weeks. Every session contains 5-10 minutes of warm-up, 5 minutes of standing exercise (站桩) with calming music, and 30-45 minutes of learning or practicing. In the first 8 sessions, 15 forms will be taught in total, averagely two forms are taught every session. In the next 8 sessions, participants will practise the complete 18-form repeatedly following the lead of an instructor with background music. Each repetition takes approximately 2 minutes 20 seconds. Apart from movements, the Taoism philosophy as the origin of Tai Chi will also be embedded during the intervention
  Interventions: Other: Tai Chi
- Control (No Intervention): Participants will be told to maintain their usual lifestyle and only attend for physical assessments

INTERVENTIONS:
Other: Dance — Exercise intervention
  Arms: Dance
Other: Tai Chi — Exercise intervention
  Arms: Tai Chi

SUMMARY:
The aim of the proposed randomised controlled study is to compare the effects and efficacy between a dance, a Tai Chi and a waiting list control group intervention over an eight-week period on physical functions and mental benefits among non-clinical adults aged between 18 and 59. The study's primary outcome is mental wellbeing and secondary parameters are physical functional and mood. A tertiary outcome will examine how the physical and mental parameters change during the learning and practice phases

DETAILED DESCRIPTION:
A double-blind, randomised controlled trial will be adopted to evaluate the effects and efficacy of an eight-week dance intervention compare with Tai Chi and control group on physical and mental benefits.

Participants will be asked to attend baseline testing one week prior to the first session, which will include lower extremity muscle strength, balance, and mental wellbeing. Participants will also be asked to fill in the mood evaluating questionnaire before and after each session to measure the acute effect of each intervention. The first four weeks of the interventions are the learning phase, participants will mainly focus on learning the movements of dance or Tai Chi. After the last session of the fourth week and before the first session of the fifth, participants will be asked to complete the previous test procedure as the mid-term test. The last four weeks are the practising phase, participants will mainly focus on practising the learned movements with reduced direction from the instructor. The post-intervention test will be completed within one week after the last session, alongside an interview on their perceptions of the intervention.

Randomisation and blinding Participants will be randomly assigned to three groups: dance, Tai Chi, and Control group, using stratified random sampling based on sex. Participant mental wellbeing scores will be ranked from highest to lowest in each sex group before being systematically assigned to one of the three intervention groups, this will reduce potential differences in baseline data between groups. All measurements will be conducted by research assistants blinded to participants' group allocation and analysis will be carried out by statistician blinded to the group and test parameters.

Interventions Participants will complete informed consent and Physical Activity Readiness Questionnaire (PAR-Q) prior to data collection. At the first testing session basic anthropometric (stature, body mass, age) and personal information (ethnicity, activity level) will be recorded and each participant issued with an Unique Identifying Code (UIC).

The Dance Group, participants will be provided with three dance genre options to choose from, ballroom dance, street dance/Hip-pop and ballet, and the most-voted genre will be delivered. Dance sessions are instructed twice a week for eight weeks. Every session lasts 45-60 minutes, containing 5-10 minutes of warm-up and 35-55 minutes of learning or practicing. In the first four weeks, a short dance sequence will be taught and in the following four weeks, participants will mainly practicing the learnt sequence along with music.

The Tai Chi Group will be given the essential 18-form of Chen's style Tai Chi Chuan which is comparatively easier for beginners to learn the iconic forms with less movements and moderate intensity. Each session lasts 45-60 minutes, twice a week for 8 weeks. Every session contains 5-10 minutes of warm-up, 5 minutes of standing exercise with calming music, and 30-45 minutes of learning or practicing. In the first 8 sessions, 15 forms will be taught in total, averaging two forms taught every session. In the following 8 sessions, participants will practise the complete 18-form repeatedly following the lead of an instructor with background music. Each repetition takes approximately 2 minutes 20 seconds. Apart from movements, the Taoism philosophy as the origin of Tai Chi will also be embedded during the intervention.

Participants in Control Group will be told to maintain their usual lifestyle and only attend for physical assessments.

The pedagogy is also considered as a vital factor in this study. Thus, instructors should record each session and briefly summarise the teaching content, descriptions, and emphases if mentioned.

Intensity monitoring and progression While delivering both dance and Tai Chi interventions, the intensity will be monitored using sessions Rate of Perceived Exertion (sRPE) using the modified Borg scale. Given the targeted age group, instructors will maintain the intended RPE between 3 (moderate) and 5 (hard), with the arbitrary unit (A.U. = RPE × session duration in minutes) from 135 to 300. Participants are asked to provide a number from CR-10 retrospectively every session and the instructor then adjusts the training load accordingly if necessary. No progression is designed in the learning phase, only studying the planned form(s) of the day. While in the practicing phase, instructors should gradually raise the standard of movements and slower the speed of practicing the full sequence to increase the difficulty and intensity.

Outcome measures The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) will be utilised to evaluate participants mental wellbeing state change. The WEMWBS is a 14-item self-evaluating scale containing hedonic and eudaimonic statements such as 'I've been feeling relaxed' or 'I've been feeling close to other people'. The respondents rate each statement spontaneously with a 5-point Likert scale from 1 to 5 (none, rarely, sometimes, often, all the time), resulting in a minimum score of 14 and maximum score of 70. The higher WEMWBS score suggests the better mental wellbeing.

The Isometric Mid-Thigh Pull (IMTP) will be used to measure lower extremity maximum strength using Hawkins Dynamic force plate. It is considered as a safe, time-effective, and reliable measurement. Participants will be asked to stand on force plates with hips and knees slightly bent. The bar height is adjusted so that it is at mid-thigh height of each participant and the height recorded. The participant grips the bar with a slight pretension. The participant is to remain completely still for 2-3 seconds before and between each repetition. The participant will then be instructed to contract as hard and as fast as possible pulling against the bar and hold the maximum pull for 2-3 seconds before resting. Each participant will carry out 3 repetitions and the maximum and mean power recorded.

The Y Balance Test (YBT) will be used to assess participants' dynamic balance. Participants will be instructed to stand barefoot unilaterally on the centre of a tape-made 'Y'. While standing on one leg, participants will reach out with their non-stance leg as far as possible in the three directions of the 'Y'. No weight can be transferred to the non-stance leg. Three attempts for each direction for each leg will be taken and calculated as a percentage of their leg length; the greatest distance for each direction will be recorded. Leg length will be measured from the greater trochanter to the lateral malleolus.

The Brunel Mood Scale (BRUMS) will be used pre and post each dance or Tai Chi session to monitor participants' mood changes. The BRUMS contains 6 categories including anger, confusion, depression, fatigue, tension, and vigour, each is comprised of 4 adjectives such as panicky, exhausted, energetic, or active. Participants are asked to indicate their mood using a 5-point Likert scale (0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely).

ELIGIBILITY:
Inclusion Criteria:

1. healthy male and female adults of any ethnicity aged from 18 to 59
2. no chronic medical conditions and
3. no physical injuries in the past 3 months that could potentially affect physical activities

Exclusion Criteria:

1. participants who are currently engaging in regular dance or Tai Chi classes
2. currently has a chronic disease or acute illness

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Well-being | Week 1, week 4 and week 8
  Warwick-Edinburgh Mental Wellbeing Scale. The total score is obtained by summing the score for each of the 14 items. The scoring range for each item is from 1 - 5 and the total score is from 14-70. Higher scores indicate greater positive mental wellbeing.

SECONDARY OUTCOMES:
Leg strength | Week 1, week 4 and week 8
  Isometric Mid-Thigh Pull: (IMTP) will be used to measure lower extremity maximum muscle strength. The participant will then be instructed to contract as hard and as fast as possible pulling against the bar and hold the maximum pull for 2-3 seconds before resting. Measurement is in kg with greater scores indicating greater muscular strength
Balance | Week 1, week 4 and week 8
  Y Balance Test: While standing on one leg, participants will reach out with their non-stance leg as far as possible in the three directions of the 'Y'. No weight can be transferred to the non-stance leg. Three attempts for each direction for each leg will be taken and calculated as a percentage of their leg length; the greatest distance for each direction will be recorded. The greater the score the better the dynamic stability/balance
Mood | 30 minutes pre and post each dance and Tai Chi intervention session up to 9 weeks
  Brunel Mood Scale (BRUMS): The acute effect of each session will be monitored. The BRUMS contains 6 categories including anger, confusion, depression, fatigue, tension, and vigour, each is comprised of 4 adjectives such as panicky, exhausted, energetic, or active. Participants are asked to indicate their mood using a 5-point Likert scale (0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely).The higher the score the more positive the mood

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wolverhampton, Walsall, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymised and then submitted to figshare account
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: available 3-months post publication for 5-years
Access Criteria: Open access promoted through publication and research centre website
URL: http://figshare.com

REFERENCES:
- [Background] Badby AJ, Mundy PD, Comfort P, Lake JP, McMahon JJ. The Validity of Hawkin Dynamics Wireless Dual Force Plates for Measuring Countermovement Jump and Drop Jump Variables. Sensors (Basel). 2023 May 17;23(10):4820. doi: 10.3390/s23104820. PMID 37430733
- [Background] Basso JC, McHale A, Ende V, Oberlin DJ, Suzuki WA. Brief, daily meditation enhances attention, memory, mood, and emotional regulation in non-experienced meditators. Behav Brain Res. 2019 Jan 1;356:208-220. doi: 10.1016/j.bbr.2018.08.023. Epub 2018 Aug 25. PMID 30153464
- [Background] Caldwell K, Harrison M, Adams M, Triplett NT. Effect of Pilates and taiji quan training on self-efficacy, sleep quality, mood, and physical performance of college students. J Bodyw Mov Ther. 2009 Apr;13(2):155-63. doi: 10.1016/j.jbmt.2007.12.001. Epub 2008 Feb 20. PMID 19329051
- [Background] Easwaran K, Gopalasingam Y, Green DD, Lach V, Melnyk JA, Wan C, Bartlett DJ. Effectiveness of Tai Chi for health promotion for adults with health conditions: a scoping review of Meta-analyses. Disabil Rehabil. 2021 Oct;43(21):2978-2989. doi: 10.1080/09638288.2020.1725916. Epub 2020 Feb 18. PMID 32070137
- [Background] Grgic J, Scapec B, Mikulic P, Pedisic Z. Test-retest reliability of isometric mid-thigh pull maximum strength assessment: a systematic review. Biol Sport. 2022 Mar;39(2):407-414. doi: 10.5114/biolsport.2022.106149. Epub 2021 Jun 1. PMID 35309521
- [Background] Haddad M, Stylianides G, Djaoui L, Dellal A, Chamari K. Session-RPE Method for Training Load Monitoring: Validity, Ecological Usefulness, and Influencing Factors. Front Neurosci. 2017 Nov 2;11:612. doi: 10.3389/fnins.2017.00612. eCollection 2017. PMID 29163016
- [Background] Koutedakis Y, Jamurtas A. The dancer as a performing athlete: physiological considerations. Sports Med. 2004;34(10):651-61. doi: 10.2165/00007256-200434100-00003. PMID 15335242
- [Background] Martin L, Oepen R, Bauer K, Nottensteiner A, Mergheim K, Gruber H, Koch SC. Creative Arts Interventions for Stress Management and Prevention-A Systematic Review. Behav Sci (Basel). 2018 Feb 22;8(2):28. doi: 10.3390/bs8020028. PMID 29470435
- [Background] Muro A, Artero N. Dance practice and well-being correlates in young women. Women Health. 2017 Nov-Dec;57(10):1193-1203. doi: 10.1080/03630242.2016.1243607. Epub 2016 Oct 4. PMID 27700698
- [Background] Nadasen K. "Life without line dancing and the other activities would be too dreadful to imagine": an increase in social activity for older women. J Women Aging. 2008;20(3-4):329-42. doi: 10.1080/08952840801985060. PMID 18983115
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Terry PC, Karageorghis CI, Curran ML, Martin OV, Parsons-Smith RL. Effects of music in exercise and sport: A meta-analytic review. Psychol Bull. 2020 Feb;146(2):91-117. doi: 10.1037/bul0000216. Epub 2019 Dec 5. PMID 31804098
- [Result] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Result] Kreutz G. Does partnered dance promote health? The case of tango Argentino. J R Soc Promot Health. 2008 Mar;128(2):79-84. doi: 10.1177/1466424007087805. PMID 18402178
- [Result] Chan AW, Yu DS, Choi KC. Effects of tai chi qigong on psychosocial well-being among hidden elderly, using elderly neighborhood volunteer approach: a pilot randomized controlled trial. Clin Interv Aging. 2017 Jan 5;12:85-96. doi: 10.2147/CIA.S124604. eCollection 2017. PMID 28115837
- [Result] Sheppard A, Broughton MC. Promoting wellbeing and health through active participation in music and dance: a systematic review. Int J Qual Stud Health Well-being. 2020 Dec;15(1):1732526. doi: 10.1080/17482631.2020.1732526. PMID 32267216
- [Result] Tao D, Gao Y, Cole A, Baker JS, Gu Y, Supriya R, Tong TK, Hu Q, Awan-Scully R. The Physiological and Psychological Benefits of Dance and its Effects on Children and Adolescents: A Systematic Review. Front Physiol. 2022 Jun 13;13:925958. doi: 10.3389/fphys.2022.925958. eCollection 2022. PMID 35770195
- Available data/document: Individual Participant Data Set — http://figshare.com — Study data will be submitted to Figshare for open science access - all identifying codes will be removed